CLINICAL TRIAL: NCT05467878
Title: The Effect of Anesthesia on Perioperative Pain Level and Analgesic Effect in Patients With Percutaneous Nephrolithotomy
Brief Title: The Effect of Anesthesia on Pain in Percutaneous Nephrolithotomy
Status: Completed | Type: Observational
Sponsor: Tugba Onur (Other Government)
Responsible Party: Sponsor-Investigator, Tugba Onur, Medical Doctor, Bursa Yuksek Ihtisas Training and Research Hospital
Organization: Bursa Yuksek Ihtisas Training and Research Hospital (Other Government)
Other Study IDs: SBÜ Bursa Hastanesi
Record Dates: First submitted 2022-04-15; First posted 2022-07-21 (Actual); Last update posted 2022-07-21 (Actual); Status verified 2022-07

CONDITIONS: Percutaneous Nephrolithotomy
Keywords: general anesthesia; postoperative pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group I: Patients undergoing regional anesthesia were studied. It can be in the form of combined spinal epidural or epidural anesthesia.
  Interventions: Other: The anesthesia and analgesia technique preferred by the anesthetist will be recorded.
- Group 2: Patients in whom general anesthesia and iv analgesic methods are preferred are in this group.
  Interventions: Other: The anesthesia and analgesia technique preferred by the anesthetist will be recorded.
- Group 3: Patients who prefer peripheral block under general anesthesia and ultrasound are in this group.
  Interventions: Other: The anesthesia and analgesia technique preferred by the anesthetist will be recorded.

INTERVENTIONS:
Other: The anesthesia and analgesia technique preferred by the anesthetist will be recorded. — In the study, the anesthesia method applied by blind anesthesiologists in the peroperative period, the drugs or techniques used for analgesia will be recorded and their effects on the postoperative period and hospital stay will be examined.There will be no intervention in the perioperative and postoperative process.

SUMMARY:
It is aimed to determine the ideal application by determining the effect of different anesthesia methods applied in percutaneous nephrolithotomy surgeries on analgesic consumption and pain level.

DETAILED DESCRIPTION:
Different anesthesia methods are used in percutaneous nephrolithotomy.In addition to traditional analgesia methods such as intravenous paracetamol, NSAIDs, opioids, various methods such as epidiural analgesia or blocks added to general anesthesia are used.In this study, it was aimed to investigate whether central or peripheral block applications are preferred in percutaneous nephrolithotomy, and the need for intraoperative and postoperative analgesics in patients.In addition, it was aimed to investigate whether there was a change in analgesic consumption, recovery and pain level, and hospital stay in patients who were given general anesthesia or regional anesthesia, in a multicentric observational manner.

ELIGIBILITY:
Inclusion Criteria:

* patient giving consent
* accessing patient information

Exclusion Criteria:

* missing information in the patient file

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 600 patients
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-01-15 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scala (VAS) | 1 days after the surgery
  Postoperative pain levels with Visual analog Scale (VAS):Between 0 and 10 points is chosen by the patients.
  0 is no pain, 10 is excessive pain.

SECONDARY OUTCOMES:
Hospital stay | after the surgery to the discharge time until 10 days
  The time elapsed from the patients to the discharge after the operation will be recorded from the files as hours.

CONTACTS AND LOCATIONS:
Overall Officials: Şeyda Efsun ŞE Özgünay, Assoc Prof, Principal Investigator — Bursa Yuksek Ihtisas Training and Research Hospital; Serra S Topal, MD, Study Chair — Bursa Yuksek Ihtisas Training and Research Hospital; Sedat S Öner, Assoc Prof, Study Chair — Bursa Yuksek Ihtisas Training and Research Hospital; Salim S Zengin, MD, Study Chair — Bursa Yuksek Ihtisas Training and Research Hospital; Şermin Ş Eminoğlu, MD, Study Chair — Bursa Yuksek Ihtisas Training and Research Hospital; Tuğba T Onur, MD, Study Chair — Bursa Yuksek Ihtisas Training and Research Hospital
Locations (1):
- Bursa YIEAH, Bursa, Yildirim, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No